CLINICAL TRIAL: NCT06802562
Title: Medical Assistance in Dying (MAiD) Requests in the Chronic Pain Clinic Setting
Brief Title: Medical Assistance in Dying Requests in Pain Clinic
Acronym: MAiD
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes MAiD Request
Record Dates: First submitted 2025-01-23; First posted 2025-01-31 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Terminal Diseases; Terminal Care; Chronic Pain; Disability or Chronic Disease Leading to Disablement
Keywords: Terminal disease; Physical disability; Chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic pain and disability.: Adult patients with chronic pain and physical disability.

SUMMARY:
Terminally ill patients often suffer existentially. Terminally ill patients with existential pain may request medical aid in dying. The Canadian government legalized Medical Assistance in Dying (MAiD) for patients unforeseeable deaths. This prospective observational study examined chronic pain clinic patients' MAiD requests. The study assessed the patients' life quality and outcomes.

DETAILED DESCRIPTION:
Adult patients diagnosed with terminal or severe intractable illnesses frequently endure existential distress. Consequently, patients with terminal illnesses who experience existential distress may contemplate or seek medical assistance in dying (MAiD). In March 2021, the Government of Canada implemented amendments to the Criminal Code to authorize Medical Assistance in Dying (MAiD) for individuals whose natural death is not reasonably foreseeable.

This prospective observational study evaluated requests made for MAiD by patients in the chronic pain clinic setting. The study assessed the quality of life and natural outcomes of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic pain and disability.

Exclusion Criteria:

* Patients without physical disability.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic pain and disability, undergoing treatment in a pain clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
How many years the patient lived after initial consultation | 3 years
  How long the patient lived naturally after the initial consultation and request for MAiD.

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD, FRCPC, Study Director — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared at the final publication.

REFERENCES:
- [Background] Bamgbade OA, Sonaike MT, Adineh-Mehr L, Bamgbade DO, Aloul ZS, Thanke CB, Thibela T, Gitonga GG, Yimam GT, Mwizero AG, Alawa FB, Kamati LO, Ralasi NP, Chansa M. Pain Management and Sociology Implications: The Sociomedical Problem of Pain Clinic Staff Harassment Caused by Chronic Pain Patients. Anesth Pain Med. 2024 May 5;14(2):e144263. doi: 10.5812/aapm-144263. eCollection 2024 Apr. PMID 39417062
- See also: Study investigator — https://orcid.org/0000-0002-8228-9260